CLINICAL TRIAL: NCT01337531
Title: Recombinant FSH Versus Highly Purified FSH in PCOS Patients Undergoing Control Ovarian Stimulation and IVF: a Prospective Randomized Study
Brief Title: Recombinant Versus Highly Purified FSH in Polycystic Ovary Syndrome (PCOS)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Genesis Center for Fertility & Human Pre-Implantation Genetics (Other)
Responsible Party: Savvas Koundouros, Responsible party is an organization
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: rFSH.- HP-FSH.PCOS
Record Dates: First submitted 2011-04-14; First posted 2011-04-19 (Estimated); Last update posted 2011-04-19 (Estimated); Status verified 2011-04

CONDITIONS: Polycystic Ovary Syndrome
Keywords: Ovarian Response in PCOS; pregnancy rate in PCOS; miscarriage rate in PCOS
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — follitropin alfa; Gonadotropins

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- gonadotropin (Experimental): recombinant or highly purified gonadotropin
  Interventions: Drug: Gonal-F, Fostimon
- Gonadotropins (Active Comparator): recombinant versus highly purified gonadotropin
  Interventions: Drug: Gonal-F, Fostimon

INTERVENTIONS:
Drug: Gonal-F, Fostimon — dosage form
  Other Names: Recombinant Gonadotropin, Highly purified Gonadotropin
  Arms: gonadotropin
Drug: Gonal-F, Fostimon — injection, daily, 10-15 days
  Other Names: Gonal-F; Fostimon
  Arms: Gonadotropins

SUMMARY:
Control ovarian stimulation responses, pregnancy and miscarriage rates are indifferent when either recombinant or highly purified follicle stimulating hormone (FSH) is used.

DETAILED DESCRIPTION:
Patients will be randomized using sealed and numbered envelopes and will be assigned to receive a similar ovarian stimulation regime incorporating either Gonal-F or highly purified Fostimon as the hormonal analog. Ovarian response using either of the two compounds, pregnancy rates and miscarriage rates will be compared to define possible statistical significance.

ELIGIBILITY:
Inclusion Criteria:

* PCOS
* Primary infertility
* No other fertility manifestation

Exclusion Criteria:

* Non PCOS
* Secondary infertility

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2011-05; Primary Completion 2011-11 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
Ovarian Response | 0-15 days post gonadotropin administration

SECONDARY OUTCOMES:
Pregnancy rate | 12-15 days post embryo replacement

CONTACTS AND LOCATIONS:
Overall Officials: Savvas N Koundouros, PhD, Principal Investigator — Genesis Center for Fertility and Human Pre-implantation Genetics
Locations (1):
- Genesis Centre for Fertility and Human Pre-implantation Genetics, Limassol, Cyprus